CLINICAL TRIAL: NCT04720222
Title: An Explorative, Monocentric, Feasibility Study to Evaluate the Detectability of the Bladder in Healthy Subjects by Ultrasound Monitoring With the Early TENA Bladder Sensor Prototype
Brief Title: Detectability of the Bladder With an Early Prototype of the Bladder Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ELECTRO; P2101 (Other: METC Number); NL76062.028.20 (Other: Central Committee on Research Involving Human Subjects)
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TENA-PROTO1 (Experimental): Investigational device. Early prototype
  Interventions: Device: TENA-PROTO1

INTERVENTIONS:
Device: TENA-PROTO1 — Each volunteer will test the TENA-PROTO1 according to a standardized protocol in multiple postural positions to evaluate the detectability of the bladder by help of the investigational device

SUMMARY:
This is an explorative, monocentric, feasibility study to evaluate the detectability of the bladder in healthy subjects by ultrasound monitoring with the early prototype of a future bladder sensor, which is intended for use for an individual suffering from urinary incontinence.

DETAILED DESCRIPTION:
The purpose of this clinical investigation with healthy subjects (defined as subjects without urological problems or lower urinary tract symptoms, assured by pre-defined inclusion and exclusion criteria) is to collect raw measurement data of the urinary bladder region of volunteers with the TENA-PROTO1, in multiple postural positions to evaluate the detectability of the bladder in the intended users and to determine the position criteria for the (future) ultrasound sensor on the lower abdomen. Secondarily, this clinical investigation aims to collect data on the adhesive and supportive belt used to fix the transducer assembly to the lower abdomen by the subject. Furthermore, safety of the subjects will be continously documented such as adverse events (AE) and device deficiencies (DD); AEs, Adverse Device Events (ADE), Severe Adverse Events (SAE), Severe Adverse Device effects (SADE), Unanticipated Serious Adverse Device Effects (USADE) and DDs.

ELIGIBILITY:
Inclusion Criteria:

* Men, women and diverse ≥ 35 and <75 years old
* Capability to understand the subject information and to provide conscious informed consent
* Signed informed consent for study participation and data protection regulations
* All subjects with childbearing potential must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of a Pearl-Index less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra uterine devices, sexual abstinence or vasectomized partner for at least 4 weeks
* Willingness to conduct a urine pregnancy test for all subjects with childbearing potential
* BMI ≥18.5 kg/m² and <40 kg/m²
* Capability and willingness to follow the following requirements: protocol, current hygiene concept and laboratory safety

Exclusion Criteria:

* Subjects with urological problems or lower urinary tract symptoms
* Subjects with breached skin, open wounds, sutures or major scar tissue in the suprapubic region.
* Subjects with active implants that can be affected by electromagnetic interference (e.g. pacemaker)
* Subjects with symptoms of constipation or diarrhea
* Subjects who are pregnant or breast feeding
* Known allergies or intolerances to one or several components of the study product
* Alcohol abuse as reported by subject and/ or suspected by investigator that impacts capability to understand the subject information and to provide conscious informed consent in the discretion of the investigator / study personnel
* Drug abuse as reported by subject and/ or suspected by investigator that impacts capability to understand the subject information and to provide conscious informed consent in the discretion of the investigator / study personnel
* Objections of the investigator to the subject's participation in the trial due to medical reasons or any other reason for which the subject should not participate in the opinion of the investigator
* Participation in any clinical investigation with systemic and/or pharmaceutical substances within the last 4 weeks and/or in parallel
* Sponsors, manufacturers or CRO staff

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Bladder detectability rate as a function of gender, BMI, age, sensor position, posture and combinations of these variables | 4 months
  Percentage of those, where the bladder was detected in total or regarding different subgroups (BMI, age, sex, postural positions and sensor location ) based on raw measurement data of the urinary bladder region of volunteers with the early prototype of the Bladder Sensor in multiple postural positions to evaluate the detectability of the bladder in the intended users
Raw measurement data for the development of an algorithm to determine the bladder filling status | 4 months
  Raw data, that has been assessed by the prototype (TENA-PROTO1) will be used to develop a product specfic algorithm (R&D outcome)

SECONDARY OUTCOMES:
Any adverse event (AE) or device deficiency (DD) | Ongoing documentation after enrolment until end of the measurement day (4 months)
  Documentation of AEs, Adverse Device Events (ADE), Severe Adverse Events (SAE), Severe Adverse Device effects (SADE), Unanticipated Serious Adverse Device Effects (USADE) and DDs.
Evaluation of the fixation methods and device regarding user needs by the subjects on a score | 4 months
  Descriptive analyses of scores assessed by a questionnaire completed by subjects regarding the adhesive and supportive belt used to fix the transducer assembly to the lower abdomen by the subject during and at the end of the measurements

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Dik, Prof., Principal Investigator — Department of Pediatric Urology, Wilhelmina Children's Hospital UMC Utrecht, P.O. Box 85090, 3508, AB, the Netherlands
Locations (1):
- Novioscan - an Essity company, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No